CLINICAL TRIAL: NCT00197522
Title: A Phase I Study Investigating Multiple Injections of Autologous CD34+ Derived Dendritic Cells Transduced With an Adenovirus Vector Expressing Inactivated HER-2/Neu in Patients With Metastatic Breast Cancer
Brief Title: Administration of Autologous Dendritic Cells (DCs) Infected With an Adenovirus Expressing Her-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Ontario Cancer Research Network (Network); Canadian Breast Cancer Research Alliance (Other); McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: file#9427-HO778-34C; CBCRA; Award # 2003HOO542
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; vaccination; dendritic cells; HER-2; CD34+ stem cells
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Biological: CD34+ derived DCs

SUMMARY:
We, the researchers at Hamilton Health Sciences, have developed a novel approach to cancer therapy using transfected dendritic cells (DCs) to generate enhanced immunity to defined tumor antigens. Dendritic cells are highly specialized antigen presenting cells found in the bone marrow, lymph nodes, skin and thymus. Infection of DCs with Adenovirus (Ad) vectors incorporating genes for defined tumor antigens enables intracellular expression and major histocompatability complex (MHC)-restricted presentation of tumor peptides by transfected DCs. Given the potent immunostimulatory properties of DCs and ability to use gene transfer to "load" DCs with tumor antigen, we hypothesize that administration of transduced autologous DCs may have potential therapeutic benefit as a cancer vaccine. We have examined Ad-tumor antigen DC based vaccination in murine models of breast cancer and melanoma. In both models, injection(s) of Ad-transduced DCs results in highly potent immune activation and antigen-specific anti-tumor responses. In these models, high levels of antigen-specific, cytotoxic effector lymphocytes that recognize and kill cancer cells directly correlates with a therapeutic response (tumor regression and/or complete protection of animals subsequently re-challenged with tumor cells). Animals demonstrating specific in vitro immunity are protected against subsequent injection of cancer cells. Moreover, we have observed complete resolution and significant long-term survival in animals with established metastatic disease with no demonstrable toxicity. As opposed to vaccination protocols with tumor peptides or purified epitopes that are MHC-I restricted (i.e. HLA-A2), we have found that injection of DCs transduced with a vector expressing the entire tumor antigen results in peptide presentation from both MHC-I and MHC-II complexes. The subsequent immune response is comprised of both CD4+ and CD8+ T cell populations. Thus, Ad-based gene transfer of tumor antigens appears to be an efficient approach: (1) enabling sustained endogenous peptide processing, and (2) facilitating DC-specific presentation to the host immune system. We have shown that using a replication deficient adenovirus vector expressing Her-2/neu DNA under the control of a human mouse mammary tumor virus (MMTV) promoter that we can transfect bone marrow derived DCs (AdHer2/DC). These cells are then used to immunize recipient mice against tumour challenge with Her2 transgenic tumour cells. The protection is antigen specific (anti Her2). On the basis of these pre-clinical studies we will initiate a pilot trial of the AdHer2/DC vaccine in Her -2/neu overexpressing patients with metastatic breast cancer. Long-term goals and implications of possible results: The goals of this initial pilot phase I study are to evaluate the safety and dosing schedule of the vaccine therapy. The vaccine will be tested in subsequent phase II and III studies to determine efficacy in comparison to standard therapies. The long-term goals are to eventually test this therapy in the adjuvant breast cancer setting in Her-2/neu overexpressing patients.

DETAILED DESCRIPTION:
Following written, informed consent, consecutive cohorts of 3-6 patients, up to a maximum of 18 patients, will be treated at increasing dose levels based on a modified Fibonacci scheme. Peripheral blood progenitor cells will be obtained from each patient following cytokine mobilization (with GM-CSF and G-CSF). Selected CD34+ cells are then cultured with human GM-CSF, human TNFα, Flt-3 ligand and human interleukin-4. The CD34+ derived dendritic cells are then transduced with an adenovirus expressing rat HER2/neu. These transduced DCs are then injected intradermally into the patient. Patients will be injected with the AdHER2/neu transduced DCs every 21 days for a total of three treatment cycles. The starting dose of dendritic cells will be 10 X 10^6 DCs. If none of the initial three patients treated at this dose experiences dose limiting toxicity (DLT) then a new cohort of three patients will be treated at a second dose level of 50 X 10^6 DCs. If any patient experiences DLT then up to six patients will be treated at the current dose level; if 2/6 or fewer patients experience DLT, we will escalate to the to the second dose level. If 3 or more patients experience DLT, the maximum tolerated dose will be deemed as exceeded and a second cohort of 3 patients will be treated at a 10 fold dose reduction of the initial dose level. The third dose level will consist of 100 x 10^6 DCs. All treatments will occur in the out-patient setting and patients will be seen prior to each injection and then monthly for at least three months following the last injection of AdHER2/neu DCs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer who are HER2/neu positive (3+ by immunohistochemistry or FISH positive) and either

  1. currently receiving hormonal therapy or are candidates for such or
  2. being considered for trastuzumab or
  3. their cancer has progressed on trastuzumab

Exclusion Criteria:

Patients are excluded from the study if they meet any one of the following criteria:

* Age less than 16 years.
* Pregnant or lactating female.
* Previous malignancy other than non-melanoma skin cancer.
* More than three prior courses of cytotoxic chemotherapy for metastatic disease.
* Concurrent use of chemotherapy, immunotherapy, or gene therapy. Concurrent hormonal therapy (tamoxifen, aromatase inhibitors or exemestane) is permitted.
* Treatment with trastuzumab within 16 weeks prior to first dose of vaccine therapy.
* Documented central nervous system metastases.
* Patients with any an acute illness that would interfere with the mobilization of stem cells or the administration of vaccination cellular therapy (ie. unstable angina, renal or liver failure, or severe chronic obstructive airways disease) are ineligible.
* Any patients requiring concurrent immunosuppressive therapy (eg. corticosteroids)
* Patients with a life expectancy of less than six months.
* ECOG performance status of >2.

Ages: 16 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2004-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and/or the maximum attainable dose (MAD) of a vaccine consisting of human autologous CD34+ DCs transduced by AdHER-2.1
To evaluate toxicity

SECONDARY OUTCOMES:
To detect evidence of clinical efficacy as measured by objective tumor reduction

CONTACTS AND LOCATIONS:
Overall Officials: Levine Mark, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada